CLINICAL TRIAL: NCT06962553
Title: Nurses' Competence and Role in Survival Prediction and Prognostic Communication: A Taboo, an Aid, or a Necessity? A Multinational Mixed- Methods Study
Brief Title: Nurses' Competence and Role in Survival Prediction and Prognostic Communication
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202501114RINE
Record Dates: First submitted 2025-04-22; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Advanced Cancer; Terminal Malignant Tumors; Hospices
Keywords: survival analysis; projections and predictions; palliative care; hospice and palliative care nursing; nurses's role

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nurses
- Doctors

SUMMARY:
[Background] Nurses' roles in survival prediction and prognostic communication have historically been limited due to role delineation, lack of formal training, and cultural norms. In Taiwan and other cultural contexts, prognostic discussions have traditionally been the purview of physicians. However, evolving paradigms in health communication, practical realities in nursing practice, and the expanded responsibilities of advanced practice nurses have highlighted the importance of nurses in this domain. Nurses frequently engage in "foreseeing" prognostic indicators through daily patient care, and emerging evidence suggests their prognostic accuracy is often comparable to or exceeds that of physicians. Despite this, the exact scope of nurses' roles in prognostication remains unclear, creating gaps in understanding the contributions, benefits, and associating factors of nurses' involvement of prognostication process.

[Aim] This mixed-methods study aims to examine hospice nurses' competencies and roles in prognostication, with a focus on their survival prediction accuracy, confidence, influencing factors, and self-perceived responsibilities.

[Method] This three-year, cross-national study adopts an explanatory sequential mixed-methods design. First, the quantitative phase utilizes a prospective cohort design, recruiting palliative nurses and physicians from ten palliative care sites across three countries. Eligible clinicians include nurses and physicians who provide care for patients with advanced cancer in palliative care settings or oncologic wards. Participating clinicians will provide weekly prognostic predictions for targeted patients and rate their confidence levels. Patients' demographic and disease-related information will also be collected to estimate survival using prediction tools. Data collection will conclude upon the patient's death or discharge. Based on the results of the quantitative phase, a descriptive qualitative study will be conducted to purposefully recruit nurses with varying levels of prediction accuracy and confidence from the quantitative phase. Semi-structured interviews will be carried out to gather qualitative data on their perspectives regarding prognostication, with a particular focus on their roles. The estimated sample size for quantitative phase is 152 nurse-physician dyads (based on 152 patients), while 20-30 nurses are expected to participate in the qualitative phase.

[Data Analysis] Descriptive statistics, area under the receiver operating characteristic (ROC) curve (AUC), Cohen's kappa, weighted kappa, McNemar's test, and ordinal logistic regression will be used to analyze quantitative data. Qualitative data will be analyzed using conventional content analysis. Nurses' Competence and Role in Survival Prediction and Prognostic Communication.

[Expecting Outcomes and Conclusion] This project uniquely highlights nurses' contributions to prognostication, aiming to generate evidence that informs future research, clinical practice, and policy development. The findings will shed light on nurses' roles, functions, potential benefits, and the barriers the face in prognostication.

ELIGIBILITY:
Inclusion Criteria:

[Inclusion criteria for patients]

* 18 years old or older
* Diagnosed with advanced solid cancer, including locally extensive or metastasis cancer
* Patients admitted to palliative care units or oncology units in the participating institutions.

[Inclusion criteria for clinicians]

* Nurses who are the primary care nurse of the included patients
* Nurses who care for the included patients for at least one shift
* Nurses who work in palliative and hospice units or team, or oncology units for over 6 months.
* Physicians who are palliative care specialists and/or physicians with palliative care trainings
* Physicians who are the primary care physician of the included patient.

Exclusion Criteria:

* Patients with hematological malignancies are excluded.
* A participated clinicians can only participate in the study up to three times, clinicians who participate in the study for more than three times are excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The research team at each site will identify eligible patients in the palliative and hospice unit and invite their physicians and nurses to participate the study.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2025-05-08 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Palliative nurses' accuracy in making survival prediction | From enrollment to the end of treatment at 2.5 years
  The results of predicted survival time estimated by participants should be specified within a range of days to weeks. The accuracy will be measured by comparing their results of prediction to: (1) the patients actual survival, (2) those of physicians, and (3) survival prediction derived from prognostic tools.
Palliative nurses' levels of confidence in making prognostic predictions | From enrollment to the end of treatment at 2.5 years
  The level of confidence will be measured on the scale of 0 to 10.

SECONDARY OUTCOMES:
Relationship between palliative nurses' demographic variables, prognostic confidence, and survival prediction accuracy | From enrollment to the end of treatment at 2.5 years
  Analysis of the association between nurses' demographic factors (e.g., age, years of experience, ward type) and their level of prognostic confidence and accuracy in predicting survival time for terminal cancer patients. Measured using structured questionnaires and comparison with actual survival outcomes.
Palliative nurses' perceptions of their roles in prognostic prediction | From enrollment to the end of treatment at 2.5 years
  Thematic analysis of interview transcripts to explore how nurses describe their roles in prognostic prediction
Themes which affect palliative nurses' prognostic prediction and level of confidence | From enrollment to the end of treatment at 2.5 years
  Identification and thematic analysis of key factors influencing palliative care nurses' prognostic predictions and their level of confidence. Themes will be derived from qualitative data collected through semi-structured and analyzed using content or thematic analysis.